CLINICAL TRIAL: NCT00162994
Title: Effect of Adenotomy and Tympanostomy on Preventing Recurrent Otitis Media in the Young Children
Brief Title: Prevention Recurrent Otitis Media in the Young Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oulu University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: K53715
Record Dates: First submitted 2005-09-10; First posted 2005-09-13 (Estimated); Last update posted 2005-12-21 (Estimated); Status verified 2002-02

CONDITIONS: Otitis Media
Keywords: recurrent otitis media; adenoidectomy; tympanostomy; young children; prevention; quality of life
MeSH Terms: conditions — Otitis Media | interventions — Adenoidectomy

INTERVENTIONS:
Procedure: adenoidectomy and tymapanostomy

SUMMARY:
The purpose of this study is to find out if young children have more benefit of the combination of adenotomy and tympanostomy than plain tympanostomy in prevention of recurrent otitis media.

DETAILED DESCRIPTION:
Recurrent otitis media is the most common bacterial disease in young children. Many risk factors are known, but benefit of operations are conflicting in children under two years of age.

In this randomized prospective controlled trial, the effect of tympanostomy tubes is compared to the effect of the combination of adenotomy and tympanostomy tubes in preventing recurrent otitis media. A control group with no active treatment is also included. The speed of recovery is studied by recording the daily symptoms and number of days of effusion comparing the differences between the groups. Life quality issues are recorded preoperatively and at about four and twelve months after the operation and are compared between the groups and to healthy children of the same age.

ELIGIBILITY:
Inclusion Criteria:

* at least 3 otitis media episodes during the last half year
* address near (< 50 km) the university hospital of Oulu

Exclusion Criteria:

* otitis media effusion lasting longer than two months without acute exacerbations
* prior adenoidectomy or tympanostomy
* head or neck malformation
* retarded child
* serious disease
* chemoprophylaxis for another disease

Ages: 10 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300
Dates: Start 2002-02; Study Completion 2005-08

PRIMARY OUTCOMES:
- number of acute otitis media
- quality of life issues

SECONDARY OUTCOMES:
- time to first recurrence
- speed of recovery of each otitis media
- number of days of middle ear effusion
- number of upper respiratory infections
- prevention of otitis media caused by pnemococcus in carrier of pneumococcus

CONTACTS AND LOCATIONS:
Overall Officials: Petri Koivunen, PhD, Study Director — Dept of Otolaryngology, University of Oulu, Finland; Olli-Pekka Alho, professor, Principal Investigator — Dept of Otolaryngology, University of Oulu, Finland; Matti Uhari, professor, Study Director — Dept of Pediatrics, University of Oulu, Finland; Tiia Kujala, MD, Principal Investigator — Dept of Otolaryngology, University of Oulu, Finland; Jukka Luotonen, PhD, Study Director — Dept of Otolaryngology, University of Oulu, Finland; Aila Kristo, MD, Principal Investigator — Dept of Otolaryngology, University of Oulu, Finland; Marjo Renko, PhD, Principal Investigator — Dept of pediatrics, University of Oulu, Finland; Tero Kontiokari, PhD, Principal Investigator — Dept of pediatrics, University of Oulu, Finland; Tytti Pokka, FK, Principal Investigator — Dept of pediatrics, University of Oulu, Finland
Locations (1):
- Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Derived] Kujala T, Alho OP, Kristo A, Uhari M, Renko M, Pokka T, Koivunen P. Quality of life after surgery for recurrent otitis media in a randomized controlled trial. Pediatr Infect Dis J. 2014 Jul;33(7):715-9. doi: 10.1097/INF.0000000000000265. PMID 24445832
- [Derived] Kujala T, Alho OP, Luotonen J, Kristo A, Uhari M, Renko M, Kontiokari T, Pokka T, Koivunen P. Tympanostomy with and without adenoidectomy for the prevention of recurrences of acute otitis media: a randomized controlled trial. Pediatr Infect Dis J. 2012 Jun;31(6):565-9. doi: 10.1097/INF.0b013e318255ddde. PMID 22466327